CLINICAL TRIAL: NCT07109154
Title: DeniLA: Comprehensive Demographics and Clinical Profile of NSCLC Patients: Analyzing Guideline-Concordant Care in First-line Treatment Patterns Observational Study (Prospective and Survey); Evaluation Patterns of Choice in First Line Treatment of Metastatic NSCLC
Brief Title: DeniLA: Comprehensive Demographics and Clinical Profile of NSCLC Patients: Analyzing Guideline-Concordant Care in First-line Treatment Patterns
Acronym: DeniLA
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133FR00224
Record Dates: First submitted 2025-07-16; First posted 2025-08-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lung Neoplasms
Keywords: Advanced Non Small Cell Lung Câncer;; Driver mutations;; PD-L1 expression;; Real World Evidence
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No

SUMMARY:
This is a prospective, observational, multicenter study, in which clinical and demographic data will be extracted from medical records. Convenience sample, with an estimated inclusion of 200 patients treated in seven participating centers.

Eligible tumors for this project will be from patients with advanced (unresectable or metastatic) non-small cell lung carcinoma, who will start first-line oncological treatment in one of the participating centers between 2025 and 2026 (between January 2025 and January 2026). Patients must be over 18 years old and data must be available in electronic medical records.

Medical records will be assessed to confirm patients' eligibility. Patients with localized disease amenable to local treatment, non-epithelial histology, small cell carcinoma and neuroendocrine tumor will not be eligible.

A survey will be designed targeting thoracic and generalist medical oncologists, aiming to understand the factors guiding the choice of first-line treatment regimens and to compare these insights with real-world data. The survey will be directed to Brazil, with an estimated of 200 filled files.

ELIGIBILITY:
Inclusion Criteria:

* Advanced (unresectable or metastatic) non-small cell lung carcinoma
* First-line oncological treatment in one of the participating centers between 2025 and 2026 (between January 2025 and January 2026)
* > 18 years old
* Data available in electronic medical records.

Exclusion Criteria:

* Localized disease amenable to local treatment
* Non-epithelial histology
* Small cell carcinoma
* Neuroendocrine tumor
* Patients with unresectable NSCLC who underwent treatment with the PACIFIC protocol and are being followed up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with advanced non-small cell lung carcinoma, treated in one of the seven centers selected, between January 2025 and January 2026.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Describe epidemiological characteristics of patients diagnosed with NSCLC in Brazil real-world. | Through study completation, an average of 2 years
  Clinical and demographic data will be extracted from medical records (gender, age at diagnosis, self-reported ethnicity, state, institutional profile (public or private), smoking status, lung cancer family history), clinical characteristics such as comorbidities, histology, extent of disease, metastasis location, tumor stage at diagnosis according AJCC eighth edition, ECOG status, frequency of biomarker and molecular testing (PDL-1 status, EGFR, ALK, ROS1, BRAF, NTRK, MET, HER2, KRAS, STK11, KEAP1). Descriptive statistics will be used to summarize the epidemiological characteristics.
Describe first-line NSCLC treatment patterns in Brazil real-world. | Through study completation, an average of 2 years
  The therapeutic choice: platinum-based therapy, ICI in monotherapy or combined, targeted therapy regimen for patients with driver mutations, TKI inhibitors, bi-specifics, ALK inhibitors, etc, will be extracted from medical records. Descriptive statistics will be used to summarize the treatment patterns.
Evaluate the concordance between the therapeutic choices and the BSCO guidelines. | Through study completation, an average of 2 years
  The concordance of real-life scenarios with the therapeutic guidelines of the Brazilian Society of Clinical Oncology (BSCO) will be assessed using Cohen's kappa coefficient.

SECONDARY OUTCOMES:
Describe of the epidemiological characteristics and first-line therapeutic patterns according all locally approved treatment approaches in NSCLC patients. | Through study completation,an average of 2 years
  The therapeutic choice on each scenario (according to EGFR, ALK, ROS1, BRAF, NTRK, MET, HER2, KRAS, STK11, KEAP1 mutations and PDL-1 status) will be collected from medical records and described on this project using descriptive statistics.
Evaluate the influence of the mutational profile and PD-L1 expression on the choice of treatment. | Through study completation, an average of 2 years
  Mutational profile and PD-L1 (presence of KRAS, KEAP1, STK11, SMARC4 co-mutations) will be collected from medical records. The influence of the mutational profile and PD-L1 expression on treatment choice will be assessed using descriptive statistics.
Evaluate the influence of clinical characteristics and mutational profile on the choice of first line treatment on EGFR mutated non-small cell lung cancer patients. | Through study completation, an average of 2 years
  The influence of clinical characteristics and mutational profile on the choice of first-line treatment for EGFR-mutated NSCLC patients (collected from medical records) will be assessed using descriptive statistics.
Evaluate differences between patterns of choice in first-line treatment between generalist medical oncologists through an online survey. | Through study completation, an average of 2 years
  Through a survey targeting thoracic and generalist medical oncologists with an estimated of 300 oncologists contacted. The differences in patterns of choice for first-line treatment among generalist medical oncologists will be summarized using descriptive statistics and compared using the Chi-squared test (or Fisher's exact test).

CONTACTS AND LOCATIONS:
Overall Officials: Clarissa Baldotto, Principal Investigator — Instituto D'Or de Pesquisa e Ensino
Locations (4):
- Brazil (4):
  - Research Site, Recife
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/